CLINICAL TRIAL: NCT00381290
Title: Intensive Diet and Exercise for Arthritis
Brief Title: Intensive Diet and Exercise for Improving Knee Osteoarthritis in Obese and Overweight Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); General Nutrition Center, Inc (Industry)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR052528 (NIH); R01AR052528 (NIH); 1R01AR052528-01A2 (NIH)
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2011-09

CONDITIONS: Osteoarthritis
Keywords: Arthritis; Arthritis, Degenerative; Knee Health; Obesity; Overweight; Osteoarthritis; Weight Loss; Diet; Exercise; Knee Pain
MeSH Terms: conditions — Osteoarthritis; Arthritis; Obesity; Overweight; Weight Loss; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Participants will follow an exercise regimen
  Interventions: Behavioral: Exercise
- 2 (Active Comparator): Participants will follow a calorie-restricted diet
  Interventions: Behavioral: Diet
- 3 (Active Comparator): Participants will follow a calorie-restricted diet and an exercise regimen
  Interventions: Behavioral: Diet; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Diet — The prescribed diet will include traditional healthy food and up to two meal replacement supplements. Initially, the diet will be set to result in an overall loss of 800 to 1000 calories per day.
  Arms: 2; 3
Behavioral: Exercise — The program will consist of 60-minute exercise sessions per week for the duration of the study. The exercise sessions will incorporate aerobic exercise and resistance training. Participants will also be encouraged to exercise at home.
  Arms: 1; 3

SUMMARY:
The purpose of this study is to compare the effects of a calorie-restricting diet, exercise, and a combination of both in reducing knee inflammation and compressive forces in obese and overweight adults with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
OA, the most common form of arthritis, occurs in about 21 million Americans. Of all the weight-bearing joints, the knee is most commonly affected by OA. Knee OA leads to physical changes to the entire joint structure, including cartilage, neighboring bone, and ligaments. Such structural changes to the knee alter joint function during movement, resulting in pain. The pain typically leads to less physical activity, leading to weight gain, followed by impaired physical function and disability.

Excessive body weight adds to the compressive forces on the knee joint and is a risk factor for OA. While there is no cure for OA, weight loss is the best nonpharmacologic way to slow OA progression. The amount of weight loss necessary to alter OA progression is unknown. The purpose of this study is to compare the effects of significant dietary restriction, exercise, and a combination of both in reducing knee inflammation and compressive forces in obese and overweight adults with knee OA. The study will also examine how diet and exercise affect everyday function and pain levels, as well as the extent of weight loss necessary for slowing OA disease progression.

This study will last 18 months. Four, 2-hour screening visits will include various questionnaires, physical exams, physical performance tests, x-rays, and blood and urine collection. Half of the participants will also undergo additional x-rays, magnetic resonance imaging (MRI), and a CT scan. Eligible participants will be randomly assigned to one of three intervention groups:

* Group 1 participants will follow a calorie-restricted diet
* Group 2 participants will follow an exercise regimen
* Group 3 participants will follow a calorie-restricted diet and an exercise regimen

Group 1 and 3 participants will aim to lose at least 10% of their body weight and drop to the next lower body mass index (BMI) class level; Group 2 participants will aim to maintain their weight. Group 1 and 3 participants will follow the prescribed diet, which will include traditional healthy food and up to two meal replacement supplements. Initially, the diet will be set to result in an overall loss of 800 to 1000 calories per day. Body weight will be monitored during weekly nutritional education and behavioral sessions. For the first 6 months, Group 1 and 3 participants will attend one individual session and three group sessions per month. During Months 7 through 18, participants will attend group sessions once every two weeks and individual sessions once every 3 months. Throughout the study, participants will record food and beverage intake in daily logs that will be collected monthly.

Group 2 and 3 participants will partake in three, 60-minute exercise sessions per week for the duration of the study. The exercise sessions will incorporate aerobic exercise and resistance training. Participants will also be encouraged to exercise at home. Body weight will be monitored monthly.

Follow-up evaluations for all participants will occur at Months 6 and 18, during which most of the screening procedures will be repeated. The Month 6 follow-up will include two study visits, and the Month 18 follow-up will include three study visits. Group 2 participants will be offered dietary counseling at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Grade II to III radiographic tibiofemoral OA of one or both knees
* Body mass index (BMI) of 27 to 37
* Sedentary lifestyle, defined as not participating in more than 30 minutes of formal exercise per week within the 6 months prior to study entry

Exclusion Criteria:

* Significant comorbidity that may pose a safety risk to the participant or otherwise interfere with the study. More information about this criterion can be found in the protocol.
* Previous acute knee injury
* Knee injection within 1 month of study entry
* Knee surgery within 6 months of study entry
* Knee OA other than tibiofemoral OA
* Unwilling or unable to change eating and physical activity habits due to environment
* Cannot speak or read English
* Excess alcohol use (21 or more drinks per week)
* Unable to finish the 18-month study or unlikely to comply with the study
* Unable to undergo MRI of the knee
* Significant cognitive impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory biomarkers | Measured at 0, 6, and 18 months (analyzed at 18 months)
Knee joint loads | Measured at 0, 6, and 18 months

SECONDARY OUTCOMES:
Bone marrow lesions | Measured at 0 and 18 months (analyzed at 18 months)
Articular cartilage | Measured at 0 and 18 months (analyzed at 18 months)
Function | Measured at 0, 6, and 18 months
Pain | Measured at 0, 6, and 18 months
Mobility | Measured at 0, 6, and 18 months
Change in quadriceps' strength and disease progression as a function of knee alignment | Measured at 0, 6, and 18 months (analyzed at 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Messier, PhD, Principal Investigator — Wake Forest University, Department of Health and Exercise Science
Locations (1):
- Wake Forest University/Wake Forest University Forest School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Focht BC, Rejeski WJ, Ambrosius WT, Katula JA, Messier SP. Exercise, self-efficacy, and mobility performance in overweight and obese older adults with knee osteoarthritis. Arthritis Rheum. 2005 Oct 15;53(5):659-65. doi: 10.1002/art.21466. PMID 16208674
- [Background] Messier SP, Gutekunst DJ, Davis C, DeVita P. Weight loss reduces knee-joint loads in overweight and obese older adults with knee osteoarthritis. Arthritis Rheum. 2005 Jul;52(7):2026-32. doi: 10.1002/art.21139. PMID 15986358
- [Background] Messier SP, Loeser RF, Miller GD, Morgan TM, Rejeski WJ, Sevick MA, Ettinger WH Jr, Pahor M, Williamson JD. Exercise and dietary weight loss in overweight and obese older adults with knee osteoarthritis: the Arthritis, Diet, and Activity Promotion Trial. Arthritis Rheum. 2004 May;50(5):1501-10. doi: 10.1002/art.20256. PMID 15146420
- [Derived] Welhaven HD, Welfley AH, Bothner B, Messier SP, Loeser RF, June RK. The metabolome of male and female individuals with knee osteoarthritis is influenced by 18-months of weight loss intervention: the IDEA trial. BMC Musculoskelet Disord. 2024 Dec 20;25(1):1057. doi: 10.1186/s12891-024-08166-7. PMID 39707277
- [Derived] Munugoda IP, Beavers DP, Wirth W, Aitken DA, Loeser RF, Miller GD, Lyles M, Carr JJ, Guermazi A, Hunter DJ, Messier SP, Eckstein F. The effect of weight loss on the progression of meniscal extrusion and size in knee osteoarthritis: a post-hoc analysis of the Intensive Diet and Exercise for Arthritis (IDEA) trial. Osteoarthritis Cartilage. 2020 Apr;28(4):410-417. doi: 10.1016/j.joca.2020.01.006. Epub 2020 Jan 31. PMID 32014493
- [Derived] Messier SP, Resnik AE, Beavers DP, Mihalko SL, Miller GD, Nicklas BJ, deVita P, Hunter DJ, Lyles MF, Eckstein F, Guermazi A, Loeser RF. Intentional Weight Loss in Overweight and Obese Patients With Knee Osteoarthritis: Is More Better? Arthritis Care Res (Hoboken). 2018 Nov;70(11):1569-1575. doi: 10.1002/acr.23608. PMID 29911741
- [Derived] Mihalko SL, Cox P, Beavers DP, Miller GD, Nicklas BJ, Lyles M, Hunter DJ, Eckstein F, Guermazi A, Loeser RF, DeVita P, Messier SP. Effect of intensive diet and exercise on self-efficacy in overweight and obese adults with knee osteoarthritis: The IDEA randomized clinical trial. Transl Behav Med. 2019 Mar 1;9(2):227-235. doi: 10.1093/tbm/iby037. PMID 29635402
- [Derived] Loeser RF, Beavers DP, Bay-Jensen AC, Karsdal MA, Nicklas BJ, Guermazi A, Hunter DJ, Messier SP. Effects of dietary weight loss with and without exercise on interstitial matrix turnover and tissue inflammation biomarkers in adults with knee osteoarthritis: the Intensive Diet and Exercise for Arthritis trial (IDEA). Osteoarthritis Cartilage. 2017 Nov;25(11):1822-1828. doi: 10.1016/j.joca.2017.07.015. Epub 2017 Jul 27. PMID 28756278
- [Derived] Beavers KM, Beavers DP, Newman JJ, Anderson AM, Loeser RF Jr, Nicklas BJ, Lyles MF, Miller GD, Mihalko SL, Messier SP. Effects of total and regional fat loss on plasma CRP and IL-6 in overweight and obese, older adults with knee osteoarthritis. Osteoarthritis Cartilage. 2015 Feb;23(2):249-56. doi: 10.1016/j.joca.2014.11.005. Epub 2014 Nov 13. PMID 25450847
- [Derived] Messier SP, Beavers DP, Loeser RF, Carr JJ, Khajanchi S, Legault C, Nicklas BJ, Hunter DJ, Devita P. Knee joint loading in knee osteoarthritis: influence of abdominal and thigh fat. Med Sci Sports Exerc. 2014 Sep;46(9):1677-83. doi: 10.1249/MSS.0000000000000293. PMID 25133996
- [Derived] Beavers DP, Beavers KM, Loeser RF, Walton NR, Lyles MF, Nicklas BJ, Shapses SA, Newman JJ, Messier SP. The independent and combined effects of intensive weight loss and exercise training on bone mineral density in overweight and obese older adults with osteoarthritis. Osteoarthritis Cartilage. 2014 Jun;22(6):726-33. doi: 10.1016/j.joca.2014.04.002. Epub 2014 Apr 15. PMID 24742955
- [Derived] Messier SP, Mihalko SL, Legault C, Miller GD, Nicklas BJ, DeVita P, Beavers DP, Hunter DJ, Lyles MF, Eckstein F, Williamson JD, Carr JJ, Guermazi A, Loeser RF. Effects of intensive diet and exercise on knee joint loads, inflammation, and clinical outcomes among overweight and obese adults with knee osteoarthritis: the IDEA randomized clinical trial. JAMA. 2013 Sep 25;310(12):1263-73. doi: 10.1001/jama.2013.277669. PMID 24065013
- [Derived] Chmelo E, Nicklas B, Davis C, Miller GD, Legault C, Messier S. Physical activity and physical function in older adults with knee osteoarthritis. J Phys Act Health. 2013 Aug;10(6):777-83. doi: 10.1123/jpah.10.6.777. Epub 2012 Oct 9. PMID 23307503
- [Derived] Messier SP, Legault C, Mihalko S, Miller GD, Loeser RF, DeVita P, Lyles M, Eckstein F, Hunter DJ, Williamson JD, Nicklas BJ. The Intensive Diet and Exercise for Arthritis (IDEA) trial: design and rationale. BMC Musculoskelet Disord. 2009 Jul 28;10:93. doi: 10.1186/1471-2474-10-93. PMID 19638215